CLINICAL TRIAL: NCT03087656
Title: Randomized Trial of Short Antibiotic Course to Decrease Post ERCP Cholangitis
Brief Title: Antibiotics to Decrease Post ERCP Cholangitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Chief Endoscopist/Associate Professor of Clinical Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-16-00880
Record Dates: First submitted 2017-03-05; First posted 2017-03-22 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Cholangitis
Keywords: levofloxacin; Ceftriaxone; Cholangitis; ERCP
MeSH Terms: conditions — Cholangitis | interventions — Ceftriaxone; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: subjects to be randomized into two arms: antibiotic arm and no antibiotic arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antibiotic arm (Active Comparator): The drugs ceftriaxone and levofloxacin will be administered to patients in the antibiotic arm.
  Interventions: Drug: Ceftriaxone; Drug: Levofloxacin
- No Antibiotic arm (No Intervention): No prophylactic antibiotics will be administered.

INTERVENTIONS:
Drug: Ceftriaxone — Intravenous Ceftriaxone will be given during the procedure.
  Other Names: Rocephin
  Arms: Antibiotic arm
Drug: Levofloxacin — Oral Levofloxacin will be given for 3 days after the procedure.
  Other Names: Levaquin
  Arms: Antibiotic arm

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an endoscopic procedure used to treat bile duct stones, obstructive jaundice, biliary leaks, and a variety of other conditions.

There is active debate whether antibiotics should be given prophylactically for ERCP outside of high risk indications including primary sclerosing cholangitis. In part this is due to a lack of appropriately powered clinical trials with adequate follow up. The aim will be to assess whether prophylactic antibiotics decrease the rate of post ERCP cholangitis as defined by the Revised Tokyo Criterion.

DETAILED DESCRIPTION:
OBJECTIVES AND PURPOSE

The aim is to determine whether a brief course of antibiotics following therapeutic ERCP can reduce post-ERCP cholangitis in patients for whom antibiotics are not already indicated.

STUDY DESIGN

The study will be a prospective, randomized trial consisting of 452 patients who are scheduled to undergo therapeutic ERCP at the LAC+USC Medical Center for standard indications. Patients undergoing ERCP for therapy of bile duct problems including choledocholithiasis, malignant obstruction, jaundice, and bile leak will be eligible. Those with mandatory antibiotic requirement will be excluded.

Patients will be randomly assigned in a 1:1 ratio using a computer generated randomization schedule and allocation will be concealed.

Patients will be randomized during the ERCP procedure, once decompression of the duct is achieved (either obstruction cleared or stent placed), to ensure that patients who are at increased risk (because of inability to decompress the duct with a stent or clearance) will be excluded from the study. Those randomized to the antibiotics arm will receive intravenous antibiotics (ceftriaxone 1gm) immediately following the ERCP procedure and will take oral antibiotics (levofloxacin 500mg) once daily for 3 subsequent days. This regimen is chosen to most closely reflect the actual clinical practice in our center. Those in the no antibiotics arm will not receive antibiotics. However, if they develop findings of cholangitis or other infection they will be treated with antibiotics. Comprehensive data including procedure indication will be recorded.

The primary outcome will be the development of post-ERCP cholangitis. Post-ERCP cholangitis will be defined by the 2013 Tokyo Guidelines

The secondary outcomes will include length of hospital stay and adverse events attributable to antibiotic use such as allergic reactions or diarrhea. All patients will be assessed 1, 3, and 7 days after the procedure by in-person visits for inpatients and telephone calls for outpatients. Patients who have fever, pain, jaundice, or signs of an adverse antibiotic outcome will be evaluated as would be done per standard clinical care.

Randomization scheme. Patients will be randomly assigned using a computer generated randomization schedule with concealed 1:1 allocation to receive a prophylactic course of antibiotics or no antibiotics.

ASSESSMENT OF EFFICACY AND SAFETY

Side effects/Toxicities to be monitored.

Major adverse outcomes which could be associated with antibiotic therapy will be recorded including unexpected allergies (such as rash or angioedema), adverse drug reactions (such as diarrhea, nausea). Patients who have diarrhea will be tested for Clostridium difficile colitis. The overall rate of these antibiotic associated events is estimated at 0.5-2%.2,13-15

CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

The outcome status (in terms of rates of cholangitis and pancreatitis as well as antibiotic toxicity and adverse events) of all eligible patients will be reported. All eligible patients who begin treatment will be included in the analysis of survival and time-to-failure.

Endpoint Definitions

Primary outcome: The primary outcome will be the development of DEFINITE post-ERCP cholangitis in <7 days.

Post-ERCP cholangitis will be defined by the 2013 Updated Tokyo Guidelines (TG13) which are the international standard.12 As the patients in this study are by definition undergoing therapeutic ERCP, criterion C will have been fulfilled.

A) Systemic Inflammation

B) Cholestasis

C) Imaging-biliary dilation and/or evidence of etiology

Secondary Outcome #1: We will compare the proportions of mild, moderate, and severe cholangitis in the two groups based on the Tokyo Guidelines (see below)12

Secondary Outcome #2: "Suspected cholangitis", as defined by the Tokyo guidelines (see table 1 above) within 7 days of ERCP.

Secondary Outcome #3: The requirement for a repeat procedure as defined by ERCP, percutaneous drainage, surgery for cholangitis within 7 days of ERCP.

Secondary Outcome #4: The length of hospital stay after ERCP.

Secondary Outcome #5: The rate of post-ERCP pancreatitis, defined as: new onset upper abdominal pain, an amylase or lipase ≥3 times the upper limit of normal, and hospitalization for ≥2 nights following ERCP.

Secondary Outcome #6: The rate of allergic reactions, serious adverse events, and C. difficile colitis attributable to antibiotic use.

The time period of all outcomes will be within 7 days of ERCP. Inpatient or telephone assessments will be done at 1, 3, and 7 days after ERCP for all patients. Any patients who are suspected to have pancreatitis or cholangitis will be advised to return to the endoscopy area immediately for a physical examination as well as vitals signs and laboratory assessment (see telephone form). In cases where there is potentially evidence of cholangitis or pancreatitis, the PI and study team will define whether the clinical constellation is most suggestive of cholangitis, pancreatitis or both processes.

STATISTICAL CONSIDERATIONS

The goal of this randomized study to determine whether a prophylactic antibiotic course can prevent cholangitis following therapeutic ERCP. Review of 200 patients at LAC USC in whom antibiotic course was given revealed a rate of cholangitis of 1%. A meta-analysis of randomized trials of antibiotics to prevent ERCP cholangitis suggested a rate of 5.8% in the control (no antibiotics group) with the largest individual trial reporting a rate of 6%.8 Pubished rates for cholangitis without antibiotics of approximately 6%. Thus at an α=0.05, β=0.8 and assuming attrition of 5% we estimate that a sample size 452 (226 per group) will be adequate to detect a statistically significant difference in the rate of post-ERCP cholangitis (assuming a difference of 1% versus 6%) within 7 days.

Intent-to-treat analyses of dichotomous outcomes will be compared using a Fischer's exact test and continuous outcomes will be compared using a Wilcoxan rank sum or T tests, depending on distribution. Multivariate logistic regression will be used for sensitivity analysis for the primary outcome if there is any imbalance in baseline characteristics, as well as if there are differential patterns of missing data or adherence between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 90 years undergoing therapeutic ERCP for standard, biliary indications including but not limited to:

  * suspected bile duct stones
  * malignant and benign biliary obstruction
  * bile leaks

Exclusion Criteria:

* Patients who are incarcerated
* Patients who are not competent to give informed consent
* Patients in whom periprocedural antibiotics are mandatory.
* These include patients with:

  * primary sclerosing cholangitis,
  * multiple biliary strictures,
  * hilar tumors,
  * neutropenia (absolute neutrophil count <500), or
  * immunosuppressive therapy.
* Patients who have been diagnosed with cholangitis or are suspected to have another active infection requiring antibiotics (such as an infected fluid collection).
* Patients who have received antibiotics within 7 days.
* Patient who have undergone ERCP within 30 days.
* Patients who undergo multiple ERCP for clinical indication will only be eligible to participate in the study for one procedure.
* Patients who have had prior biliary surgeries.
* Patients in whom bile duct decompression is unsuccessful will be excluded as these patients are at increased risk of cholangitis.
* Patients with immediate procedural complications such as a bowel perforation.
* Patients undergoing ERCP for diagnostic purposes only will be excluded as the aim is to study the role of antibiotics in those undergoing therapeutic ERCP.
* Pregnant women
* Patient with allergies to fluoroquinolones. Patient with allergies to cephalosporins or penicillin's may receive fluoroquinolones if they are randomized to antibiotics arm.
* Patients with renal insufficiency (creatinine clearance <80ml50ml/minute), in whom dose modifications are necessary.

Withdrawal Criteria:

* Patients who withdraw consent will be withdrawn from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2024-02-23 (Estimated); Study Completion 2024-02-23 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who develop Post-ERCP Cholangitis as defined by the revised Tokyo criterion. | 1 week
  The primary outcome will be the proportion of patients who develop develop post-ERCP cholangitis as defined by the Revised Tokyo criterion within 1 week of ERCP.

SECONDARY OUTCOMES:
Days of hospitalization | 1 week
  The number of days of hospitalization following ERCP will be compared among the two groups.
Proportion of patients who develop adverse events of antibiotics | 1 week
  The proportion of patients in the two groups who develop allergic reactions, C. difficile colitis, and other adverse symptoms attributable to antibiotic use will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, Principal Investigator — University of Southern California Health Science Center
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sauter G, Grabein B, Huber G, Mannes GA, Ruckdeschel G, Sauerbruch T. Antibiotic prophylaxis of infectious complications with endoscopic retrograde cholangiopancreatography. A randomized controlled study. Endoscopy. 1990 Jul;22(4):164-7. doi: 10.1055/s-2007-1012830. PMID 2209498
- [Result] van den Hazel SJ, Speelman P, Dankert J, Huibregtse K, Tytgat GN, van Leeuwen DJ. Piperacillin to prevent cholangitis after endoscopic retrograde cholangiopancreatography. A randomized, controlled trial. Ann Intern Med. 1996 Sep 15;125(6):442-7. doi: 10.7326/0003-4819-125-6-199609150-00002. PMID 8779455
- [Result] Glomsaker T, Soreide K, Hoff G, Aabakken L, Soreide JA; Norwegian Gastronet ERCP group. Contemporary use of endoscopic retrograde cholangiopancreatography (ERCP): a Norwegian prospective, multicenter study. Scand J Gastroenterol. 2011 Sep;46(9):1144-51. doi: 10.3109/00365521.2011.594085. Epub 2011 Jun 22. PMID 21692712
- [Result] Cotton PB, Garrow DA, Gallagher J, Romagnuolo J. Risk factors for complications after ERCP: a multivariate analysis of 11,497 procedures over 12 years. Gastrointest Endosc. 2009 Jul;70(1):80-8. doi: 10.1016/j.gie.2008.10.039. Epub 2009 Mar 14. PMID 19286178
- [Result] Christensen M, Matzen P, Schulze S, Rosenberg J. Complications of ERCP: a prospective study. Gastrointest Endosc. 2004 Nov;60(5):721-31. doi: 10.1016/s0016-5107(04)02169-8. PMID 15557948
- [Result] Andriulli A, Loperfido S, Napolitano G, Niro G, Valvano MR, Spirito F, Pilotto A, Forlano R. Incidence rates of post-ERCP complications: a systematic survey of prospective studies. Am J Gastroenterol. 2007 Aug;102(8):1781-8. doi: 10.1111/j.1572-0241.2007.01279.x. Epub 2007 May 17. PMID 17509029
- [Result] Bodger K, Bowering K, Sarkar S, Thompson E, Pearson MG. All-cause mortality after first ERCP in England: clinically guided analysis of hospital episode statistics with linkage to registry of death. Gastrointest Endosc. 2011 Oct;74(4):825-33. doi: 10.1016/j.gie.2011.06.007. Epub 2011 Aug 11. PMID 21835401
- [Result] Bai Y, Gao F, Gao J, Zou DW, Li ZS. Prophylactic antibiotics cannot prevent endoscopic retrograde cholangiopancreatography-induced cholangitis: a meta-analysis. Pancreas. 2009 Mar;38(2):126-30. doi: 10.1097/MPA.0b013e318189fl6d. PMID 19238021
- [Result] ASGE Standards of Practice Committee; Khashab MA, Chithadi KV, Acosta RD, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Faulx AL, Fonkalsrud L, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Shaukat A, Wang A, Cash BD. Antibiotic prophylaxis for GI endoscopy. Gastrointest Endosc. 2015 Jan;81(1):81-9. doi: 10.1016/j.gie.2014.08.008. Epub 2014 Nov 11. No abstract available. PMID 25442089
- [Result] Cotton PB, Connor P, Rawls E, Romagnuolo J. Infection after ERCP, and antibiotic prophylaxis: a sequential quality-improvement approach over 11 years. Gastrointest Endosc. 2008 Mar;67(3):471-5. doi: 10.1016/j.gie.2007.06.065. Epub 2007 Dec 3. PMID 18061594
- [Result] Brand M, Bizos D, O'Farrell P Jr. Antibiotic prophylaxis for patients undergoing elective endoscopic retrograde cholangiopancreatography. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD007345. doi: 10.1002/14651858.CD007345.pub2. PMID 20927758
- [Result] Kiriyama S, Takada T, Strasberg SM, Solomkin JS, Mayumi T, Pitt HA, Gouma DJ, Garden OJ, Buchler MW, Yokoe M, Kimura Y, Tsuyuguchi T, Itoi T, Yoshida M, Miura F, Yamashita Y, Okamoto K, Gabata T, Hata J, Higuchi R, Windsor JA, Bornman PC, Fan ST, Singh H, de Santibanes E, Gomi H, Kusachi S, Murata A, Chen XP, Jagannath P, Lee S, Padbury R, Chen MF, Dervenis C, Chan AC, Supe AN, Liau KH, Kim MH, Kim SW; Tokyo Guidelines Revision Committee. TG13 guidelines for diagnosis and severity grading of acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2013 Jan;20(1):24-34. doi: 10.1007/s00534-012-0561-3. PMID 23307001
- [Result] Carignan A, Allard C, Pepin J, Cossette B, Nault V, Valiquette L. Risk of Clostridium difficile infection after perioperative antibacterial prophylaxis before and during an outbreak of infection due to a hypervirulent strain. Clin Infect Dis. 2008 Jun 15;46(12):1838-43. doi: 10.1086/588291. PMID 18462108
- [Result] Johannes CB, Ziyadeh N, Seeger JD, Tucker E, Reiter C, Faich G. Incidence of allergic reactions associated with antibacterial use in a large, managed care organisation. Drug Saf. 2007;30(8):705-13. doi: 10.2165/00002018-200730080-00007. PMID 17696583